CLINICAL TRIAL: NCT05278455
Title: Smartphone-Delivered Lifestyle Medicine Intervention for Generalized Anxiety Symptoms: A Randomized Controlled Trial
Brief Title: Self-help Lifestyle Medicine for Generalized Anxiety Symptoms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Fiona YY Ho, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PSY020
Record Dates: First submitted 2022-03-04; First posted 2022-03-14 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Generalised Anxiety Disorder
Keywords: Generalised anxiety disorder; Smartphone-based; Multicomponent lifestyle medicine intervention; Self-help; Randomised controlled trial
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle Medicine Group (Experimental): Lifestyle medicine smartphone app The lifestyle medicine app contains eight weekly modules that cover healthy eating, exercise, stress management, sleep management, lifestyle psychoeducation, and goal setting.
  Interventions: Behavioral: Lifestyle Medicine
- Waitlist Control Group (No Intervention): The waitlist control group will receive access to the lifestyle medicine app at the end of the study.

INTERVENTIONS:
Behavioral: Lifestyle Medicine — A smartphone-delivered application with a series of lifestyle medicine components, including lifestyle psychoeducational, physical activity, dietary recommendations, stress management, sleep management, and motivation and goal-setting techniques.
  Arms: Lifestyle Medicine Group

SUMMARY:
This study will examine the effects of smartphone-based lifestyle medicine for alleviating generalised anxiety symptoms in Chinese population. Since a range of lifestyle factors are involved in the pathogenesis and progression of generalised anxiety disorder ( Cox & Olatunji, 2016; Dale et al., 2014; Vøllestad et al., 2012), modifying different lifestyle factors simultaneously, for examples, diet, exercise, stress and sleep, may be effective to reduce generalised anxiety symptoms. Recent studies indicate that service users are showing an increasing interest in self-help interventions for common mental disorders because of their accessibility and low cost (Marshall et al., 2021; Weisel et al., 2019). Nonetheless, to date, only limited self-help interventions that target lifestyle medicine for generalised anxiety symptoms are available.

This study will be a randomised controlled trial on the effects of a self-help smartphone-based lifestyle medicine intervention for reducing generalised anxiety symptoms in Chinese population. Prior to all study procedures, eligible participants will be required to complete an online informed consent (with telephone support). Around 50 eligible participants will be randomly assigned to either smartphone-based lifestyle medicine (LM group) or the waitlist control group (WL group) in a ratio of 1:1. The randomization will be performed by an independent assessor using a computer-generated list of numbers. Participants in the LM group will receive the multicomponent lifestyle medicine intervention via the app for 8 weeks, whilst the WL control group will receive the intervention after trial completion. The primary outcomes will be the level of generalised anxiety symptoms at immediate and 3-month post-intervention assessments; while the secondary outcomes will be the level of depressive symptoms, insomnia symptoms, physical activity, health-related quality of life, functional impairment, health-promoting behaviours, and intervention acceptability at immediate and 3-month post-intervention assessments.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong residents
* Aged ≥ 18 years
* Have a Generalized Anxiety Disorder-7 (GAD-7) score ≥ 8
* Able to read Chinese and type in Chinese or English
* Have an Internet-enabled mobile device (iOS or Android operating system)
* Willing to provide informed consent and comply with the trial protocol

Exclusion Criteria:

* Current involvement in psychotherapy or recent changes in medication for anxiety
* A Patient Health Questionnaire-9 (PHQ-9) item 9 score > 2, indicating a serious level of suicidal risk (referral information to professional mental health services will be provided)
* Self-disclosure of having unsafe health conditions for which physical activity or a change in diet was contraindicated by physicians
* Self-disclosure of a diagnosis of any major psychiatric, medical or neurocognitive disorders that make participation unsuitable or that may interfere with the adherence to the lifestyle modifications

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Change in the Generalized Anxiety Disorder-7 (GAD-7) | Baseline, immediate post-intervention, and 3-month post-intervention
  GAD-7 is a seven-item scale for assessing the level of generalized anxiety in the past two weeks. It comprises questions related to feelings of anxious and worry in daily lives. This four-point Likert scale is rated from 0 (not at all) to 3 (almost everyday), and the cut off score on the sum of each item will be the standard to differentiate the anxiety level (5, 10, 15 correspond to mild, moderate and severe respectively)

SECONDARY OUTCOMES:
Change in the Patient Health Questionnaire (PHQ-9) | Baseline, immediate post-intervention, and 3-month post-intervention
  PHQ-9 is a nine-item scale for assessing the level of depressive symptoms in the past two weeks. This four-point Likert scale is rated from 0 (not at all) to 3 (almost every day), and the cut off scores on the sum of each item will be the standard to differentiate the depressive level (5, 10, 15, 20 correspond to mild, moderate, moderately severe and severe respectively)
Change in the Insomnia Severity Index (ISI) | Baseline, immediate post-intervention, and 3-month post-intervention
  ISI is a seven-item scale for measuring the severity of sleep disturbance. This five-point Likert scale is rated from 0 to 4 for each item, and a higher total score indicates the more severe of the insomnia condition (8, 15, 22 correspond to subthreshold insomnia, moderate clinical insomnia and severe clinical insomnia respectively).
Change in the Short Form (Six-Dimension) Health Survey (SF-6D) | Baseline, immediate post-intervention, and 3-month post-intervention
  SF-6D is a single index and preference-based questionnaire for measuring individual's quality of lives in the following six domains, including physical functioning, role limitation, social functioning, bodily pain, mental health, and vitality.
Change in the Health-Promoting Lifestyle Profile (HPLP II) | Baseline, immediate post-intervention, and 3-month post-intervention
  HPLP-II is a 52-item questionnaire for measuring the present lifestyle or personal habits with six sub-scale domains, including health responsibility, physical activity, nutrition, spiritual growth, interpersonal relations, and stress management. The inventory uses a four-point Likert scale, from 1 (never) to 4 (routinely), to evaluate the frequency of items asked to the participants.
Change in the Sheehan Disability Scale (SDS) | Baseline, immediate post-intervention, and 3-month post-intervention
  SDS is a three-item, self-reported 10-point visual analog scale on measuring one's severity level of impairment on three dimensions, including work/school, social life, and family life.
Change in the Credibility-Expectancy Questionnaire (CEQ) | Baseline and immediate post-intervention
  CEQ is a self-reported 6-item inventory for assessing one's attitude towards the credibility and expectancy of the intervention contents.
Change in the Treatment Acceptance Questionnaire (TAQ) | Baseline and immediate post-intervention
  TAQ is a self-reported, six-item questionnaire that is rated by a seven-point Likert scale from 1 to 7, and it aims at evaluating the clients' attitude toward the treatment sessions by six domains, including acceptability, ethics, effectiveness, negative side effects, the therapist's knowledge, and the therapist's trustworthiness.
Change in the International Physical Activities Questionnaire-Chinese version (IPAQ-C) | Baseline, immediate post-intervention, and 3-month post-intervention
  IPAQ-C is a 5-item questionnaire that measures the amount of sitting time, walking time, and moderate and vigorous exercise during the last 7 days. Different exercise types are categorized and rated as different metabolic equivalent tasks, while a higher score of the sum of total items represents a higher intense of activity level.

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Shatin, Hong Kong